CLINICAL TRIAL: NCT06845384
Title: Registry of Acute Coronary Syndrome in the Regional Cardiovascular Center
Acronym: STOCS
Status: Active, not recruiting | Type: Observational
Sponsor: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Collaborators: Stupino Clinical Hospital, Moscow Region State Medical Institution (Unknown)
Responsible Party: Sponsor
Other Study IDs: 03-06/24
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Аcute Coronary Syndrome
Keywords: acute coronary syndrome; percutaneous coronary intervention; unstable angina; acute myocardial infarction
MeSH Terms: conditions — Acute Coronary Syndrome; Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No

SUMMARY:
The study is a prospective registry of patients consequently admitted to the regional cardiovascular center with a diagnosis of acute coronary syndrome, in order to study the behavior of patients from the first minutes of the onset of the anginal syndrome, and influence of the delay in calling of ambulance on short-term and long-term outcomes of the disease. Other factors which may influence short-term and long-term outcomes will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 and over, permanently residing in the Moscow region and in Moscow.
2. Patients hospitalized in the Regional Vascular Center of Stupino Clinical Hospital (GBUZ MO SKB) with a diagnosis of ACS with and without ST-segment elevation.
3. Signing an informed consent form to participate in the study and the processing of personal data, as well as conducting a telephone survey during the follow-up.

Exclusion Criteria:

1. The patient's refusal to participate in the study and to allow the use of personal data during the study.
2. The presence of mental illness.
3. The patient plans to leave Russia for permanent or long-term residence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients consequently admitted to the regional cardiovascular center with a diagnosis of acute coronary syndrome, in order to study the behavior of patients from the first minutes of the onset of the anginal syndrome, and influence of the delay in calling of ambulance on short-term and long-term outcomes of the disease.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | 1 year and 3 years

SECONDARY OUTCOMES:
Сombined secondary end-point | 1 year and 3 years
  Rate of nonfatal myocardial infarction, nonfatal stroke, hospitalization for decompensated heart failure, and emergency invasive cardiac interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Martsevich, D.M., professor, Study Director — National Medical Research Centre for Therapy and Preventive Medicine, Moscow, Russia
Locations (1):
- National Medical Research Centre for Therapy and Preventive Medicine, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No